CLINICAL TRIAL: NCT00002041
Title: Evaluation of Amphotericin B in the Treatment of Biopsy Proven Candida Esophagitis in Immunocompromised Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001A; 875-10
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: Candidiasis, Esophageal; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Esophagitis; Acquired Immunodeficiency Syndrome; Amphotericin B; Candidiasis, Oral
MeSH Terms: conditions — Candidiasis; HIV Infections; AIDS-Related Opportunistic Infections; Esophagitis; Acquired Immunodeficiency Syndrome; Candidiasis, Oral | interventions — Amphotericin B

INTERVENTIONS:
Drug: Amphotericin B

SUMMARY:
To determine the appropriate duration of amphotericin B therapy for Candida esophagitis. To compare the effectiveness of two different amphotericin B doses in the treatment of biopsy-proven Candida esophagitis. To determine if low-dose amphotericin B is less toxic than standard dose therapy during a limited treatment period. To evaluate pharmacokinetic and pharmacodynamic parameters of the two different dosing regimens.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with histological or clinical (skin rash, cotton wool exudates, Candida endophthalmitis, etc.) evidence of disseminated candidiasis are excluded.

Concurrent Medication:

Excluded:

* Systemic administration of amphotericin B for a proven or suspected systemic fungal infection.

Patients with the following are excluded:

* Documented Candida fungemia.
* Histological or clinical (skin rash, cotton wool exudates, Candida endophthalmitis, etc.) evidence of disseminated candidiasis.
* Systemic administration of amphotericin B for a proven or suspected systemic fungal infection.
* Patient refusal to enter study.

Patient must be an immunosuppressed host, with biopsy-proven Candida esophagitis.

* Patients with polymicrobial esophagitis will be included as long as Candida esophagitis is documented by esophageal biopsy.
* Informed consent must be signed and obtained.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Bristol - Myers Squibb Co, Princeton, New Jersey, United States